CLINICAL TRIAL: NCT04517448
Title: Quality of Life of Patients Over 75 Yars Undergoing Palliative Chemotherapy for Digestive Cancer
Brief Title: Quality of Life of Patients Over 75 Yars Undergoing Palliative Chemotherapy
Acronym: EQLVCPAL
Status: Terminated | Type: Observational
Why Stopped: End of recruitment - Number of required subjects enrolled
Sponsor: Centre Hospitalier de la côte Basque (Other)
Responsible Party: Principal Investigator, AUDEMAR Franck, Principal investigator, Centre Hospitalier de la côte Basque
Other Study IDs: P-2020/01
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Pancreatic Cancer; Biliary Cancer; Hepatic Cancer; Oesophageal Cancer; Gastric Cancer
Keywords: Digestive cancer, age other 75 years old, palliative therapy, quality of life
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms; Liver Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this research is to evaluate the quality of life of patients over 75 years of age undergoing palliative chemotherapy for digestive cancer. It is a non-interventional study that evaluates the quality of life before and after a cycle of chemotherapy with a composite criterion including: a standardized questionnaire "Cancer specific quality of Life questionnaire" (QLQC30), an assessment of autonomy by "Activity of daily living" questionnaire (ADL), and the number of days of hospitalization.

DETAILED DESCRIPTION:
The number of patients undergoing chemotherapy continues to increase as well as the age of cancer patients, it is estimated that in 2050 one cancer out of two will be discovered in a person over 75 years of age. Digestive cancers account for the majority of these patients, the goals of these palliative chemotherapies are to improve survival and maintain or improve quality of life. Since the 2009 cancer plan, a specific geriatric onco-geriatrics organization has been set up with the creation of geriatric onco-coordination units. One of the objectives of this plan is to achieve a 5% inclusion rate of patients over 75 years of age in clinical trials. However, there are relatively few studies in patients over 75 years of age concerning quality of life, as they are often excluded from trials and survival is preferred as the primary outcome. This observational study evaluates the quality of life of patients at the time of the first chemotherapy treatment and then at the end of the first cycle of chemotherapy at 3 months by a standardized questionnaire, an evaluation of autonomy and the number of days of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age over 75 years old
* Suffering from digestive cancer : colorectal, pancreatic, biliary, oesophageal, gastric
* Palliative cancer : not resectable, multimetastatic
* Decision in multi-disciplinary liaising meeting (CPR) to perform a first course of palliative chemotherapy
* Having received an informed consent form
* Understanding french language

Exclusion Criteria:

* Cognitive disorders
* Patient benefiting from a legal protection measure
* Life expectancy below 1 year
* Not understanding french language

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Patient other 75 years old, undergoing a palliative chemotherapy for a digestive cancer : colorectal, pancreatic, biliary, oesophageal, gastric, proved by histology, whatever the histologic type (adenocarcinoma, epidermoid carcinoma, neuroendocrine carcinoma); at a palliative stage (not resecable, multimetastatic) and who will perform a first course of palliative chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Change in the response scores to the standardized questionnaire Quality of life questionnaire in cancer patient | Before first chemotherapy and at Month 3 of chemotherapy
  The primary outcome is a composite criterion comparing the response scores to the standardized questionnaire Quality of life in cancer patient . These data will be collected during the first inpatient chemotherapy course in hospitalization and during the last chemotherapy before evaluation. A higher score would mean a worsening of the situation

SECONDARY OUTCOMES:
Change in the Activity of daily living score | Before first chemotherapy and at Month 3 of chemotherapy
  The secondary outcome in to compare the Activity of daily living score at first chemotherapy and at the end of the first cycle at 3 months. We will collect the patient's place of residence in order to look for possible institutionalization, which is an important marker of quality of life. A higher score would mean a worsening of the situation.

CONTACTS AND LOCATIONS:
Locations (1):
- CH Côte Basque, Bayonne, France